CLINICAL TRIAL: NCT03101709
Title: The Safety and Efficacy of CART-19 Cells in Relapse and Refractory Patients With CD19+ B-cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: The Beijing Pregene Science and Technology Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH109
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Cyclophosphamide; fludarabine; CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART-19 (Experimental): patients will receive a pre-conditioning with cyclophosphamide and fludarabine before infusion of CART-19 cells. The CART-19 cells are to be administered on day0,day1,day2.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: CART-19

INTERVENTIONS:
Drug: Cyclophosphamide — patients will receive a standard pre-conditioning regime with cyclophosphamide 0.8-1.0g/m2/day IV for 2 days(Day-5 to day-4).
Drug: Fludarabine — Fludarabine 25 mg/m2/day IV for 3 days (Day-5 to day-3).
Biological: CART-19 — CART-19 cells will be administered using a split dose on day0(10%), 1(30%), and 2(60%) after completion of the chemotherapy.

SUMMARY:
This is a clinical study to observe the safety and feasibility of chimeric antigen receptor 19 (CART-19) cells in relapsed and refractory patients with CD19+ B cell lymphoma.

DETAILED DESCRIPTION:
This is a study for the patients with B cell lymphoma. Subjects will be staged and the suitability of their T cells for CART-19 manufacturing will be determined at entry phase. Subjects will be collected their T cells and modify them, the modification is a genetic change, that CD19:4-1BB:CD3 modified T cells, in order to tells the T cells to recognize their target tumor cells and potentially kill them, but not other normal cells in the subject's body. The CART cells will then be expanded in vitro and then administered to subjects.

The purpose of this study is to assess ssess the safety and feasibility of CART-19 cells in the patients with relapsed and refractory CD19+ B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 70 years, expected survival > 3 months;
2. CD19 positive B-cell lymphoma;
3. KPS >80;
4. Having at least one measurable lesions;
5. Cardiac function: 1-2 levels; Liver: TBIL≤3ULN，AST ≤2.5ULN，ALT ≤2.5ULN; kidney: Cr≤1.25ULN; bone marrow: WBC ≥ 3.0×109/L, Hb ≥90 g/L, PLT ≥ 80×109/L）;
6. No serious allergic constitution;
7. No other serous diseases that conflicts with the clinical program;
8. No other cancer history;
9. No serious mental disorder;
10. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. Pregnant or lactating women; (female participants of reproductive potential must have a negative serum or urine pregnancy test);
2. Uncontrolled active infection, HIV infection, syphilis serology reaction positive;
3. Active hepatitis B or hepatitis C infection;
4. Recent or current use of glucocorticoid or other immunosuppressor;
5. With severe cardiac, liver, renal insufficiency, diabetes and other diseases;
6. Transaminase >2.5ULN, Bilirubin >3ULN，Creatinine>1.25ULN
7. Participate in other clinical research in the past three months; previously treatment with any gene therapy products;
8. Researchers think of that does not fit to participate in the study, or other cases that affect the clinical trial results;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
safety as assessed by the occurence of study related adverse events | 6 months
  monitor the occurence of study related adverse events

SECONDARY OUTCOMES:
efficacy assessed by anti-tumor activity of CART-19 cells | 2 years
  anti-tumor activity of CART-19 cells will be determined in a follow-on study
duration of CART-19 | 2 years
  Determine duration of in vivo survival of CART-19 cells

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China